CLINICAL TRIAL: NCT03373162
Title: Measuring the Functional Effects of Botox on the Brain Using MR Spectroscopy and fMRI
Brief Title: Functional Effects of Botox on the Brain Using MRS and fMRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-3377
Record Dates: First submitted 2017-10-02; First posted 2017-12-14 (Actual); Results first posted 2019-04-26 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Healthy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRI Scans Pre and Post-Botox Injection (Experimental): Participants will receive MRI scans pre and post-Botox injection, including magnetic resonance spectroscopy, structural, and functional MRI.
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — This study is a pre- and post-design. One scan will be collected prior to BOTOX injection and the second will be collected 14-21 days post-injection. BOTOX injections will be limited to 20 units in the glabellar area, as approved by the FDA .
  Other Names: Botox

SUMMARY:
The injection of BOTOX into peripheral muscles has been shown to have therapeutic effects in a growing number of indications including disorders involving skeletal muscle (e.g., strabismus, blepharospasm, cervical dystonia, spasticity, cosmetic), smooth muscle (e.g., bladder), glands (axillary hyperhidrosis) and nociceptive pain (e.g. migraine) (Brin. 2014). Recently, several studies have suggested that peripheral BOTOX injections in the region of the glabellar lines (muscles around the eyes) may be effective in treating major depression and chronic migraine. However, the mechanism underlying the effect of peripheral BOTOX injections on the brain is not well understood. Therefore, the Investigators propose to further explore the functional effects of BOTOX injections on brain in healthy controls. The approach will involve the measurement of brain metabolites in the brainstem using MRS as well as an investigation of the functioning and connectivity between regions of the brain using resting state MRI and high resolution fMRI.

DETAILED DESCRIPTION:
Participants will receive one MRI scan session prior to a standardized, clinical dose of BOTOX injected into the forehead per FDA-approved procedures. Participants will then undergo a second MRI scan session 2-3 weeks later, after the BOTOX has taken maximal effect. Examining fMRI of the brainstem and the functional connectivity of the brainstem and connections to cortex, may provide additional insight into the effects of BOTOX on neurologic and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Ages 30-40 years of age
* Right-handed
* Normal or corrected-to-normal vision
* No history of psychiatric, neurological, or medical co-morbidities that might interfere with normal brain functioning
* Fluent in English
* Moderate to severe glabellar lines

Exclusion Criteria:

* Pregnancy
* Ferrous metal, a pacemaker, or other battery-operated device implanted in the body
* Claustrophobia
* Known hypersensitivity to Botulinum Toxin
* Infection on the forehead or between the eyes
* Urinary tract infection

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Stark, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stark S, Stark C, Wong B, Brin MF. Modulation of amygdala activity for emotional faces due to botulinum toxin type A injections that prevent frowning. Sci Rep. 2023 Feb 27;13(1):3333. doi: 10.1038/s41598-023-29280-x. PMID 36849797

RESULTS

PARTICIPANT FLOW:
Groups:
- MRI Scans Pre and Post-Botox Injections: Participants will receive MRI scans pre and post-Botox injection
  onabotulinumtoxinA: This study is a pre- and post-design. One scan will be collected prior to BOTOX injection and the second will be collected 14-21 days post-injection. BOTOX injections will be limited to 20 units in the glabellar area, as approved by the FDA .
Period: Overall Study
Arm/Group | MRI Scans Pre and Post-Botox Injections
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-Post: Participants will receive MRI scans pre and post-Botox injection
  onabotulinumtoxinA: This study is a pre- and post-design. One scan will be collected prior to BOTOX injection and the second will be collected 14-21 days post-injection. BOTOX injections will be limited to 20 units in the glabellar area, as approved by the FDA .
Arm/Group | Pre-Post
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
MRS measures of Glx normalized to Creatine [Mean (Standard Deviation); unit: Concentration Ratio] | 1.9 (.49)
BOLD fMRI activity in Left Amygdala: Happy faces vs baselines task [Mean (Standard Deviation); unit: Beta value] | 1.4 (.06)
BOLD fMRI activity in Left Amygdala: Angry faces vs baselines task [Mean (Standard Deviation); unit: Beta values] | .08 (.08)

OUTCOME MEASURES:

1. Primary Outcome: Glutamate + Glutamine (Glx)/Creatine Ratio as Measured by MRS in the Brainstem Pre and Post-Botox
Description: Determine whether there are metabolic differences in the brain stem in healthy individuals as a result of BOTOX using MRS. Participants were scanned 1-13 days prior to Botox injections in the glabellar region and then again 14-21 days post-injection when the Botox had reached effectiveness. Metabolite FIDs were averaged within each task and processed using TARQUIN (v.4.3.6) software for spectral fitting. The acquired MRS spectra was corrected for tissue type and T2 relaxation differences. Using TARQUIN we obtained values for Glutamate + Glutamine (Glx), normalized by Creatine.
Time Frame: 15-33 days between pre and post-Botox scans
Measure: Mean (Standard Error); unit: Brainstem GLX/Cr
Groups:
- MRI Scans Pre and Post-Botox Injection: Participants will receive MRI scans pre and post-Botox injection
  onabotulinumtoxinA: This study is a pre- and post-design. One scan will be collected prior to BOTOX injection and the second will be collected 14-21 days post-injection. BOTOX injections will be limited to 20 units in the glabellar area, as approved by the FDA .
Arm/Group | MRI Scans Pre and Post-Botox Injection
Number analyzed (Participants) | 10
Brainstem GLX/Cr | .12 (.44)

2. Primary Outcome: Change From Baseline in Functional MRI Mean Blood Oxygen Level Dependent (BOLD) Response in the Amygdala
Description: Understand the effect of BOTOX on functional activity (measured using fMRI) in the brain. Participants were scanned 1-13 days prior to Botox injections in the glabellar region and then again 14-21 days post-injection when the Botox had reached effectiveness. Participants viewed Happy and Angry faces and rated each one as pleasant or unpleasant. We then masked activity in the amygdala to investigate the difference in BOLD response for collapsed across emotion following Botox injections.
Time Frame: 15-33 days between pre and post-Botox scans
Measure: Mean (Standard Error); unit: fMRI BOLD in Left Amygdala
Arm/Group | MRI Scans Pre and Post-Botox Injection
Number analyzed (Participants) | 10
fMRI BOLD in Left Amygdala | -1.7 (.45)

3. Secondary Outcome: Number of Participants With Structural Brain Volume Change Following Botox Injections
Description: Participants were scanned 1-13 days prior to Botox injections in the glabellar region and then again 14-21 days post-injection when the Botox had reached effectiveness. Structural scans for each participant were segmented using Freesurfer's automatic software for volumetric measures and then normalized by dividing by total intracranial volume for each participant. We then conducted t-tests for pre- vs. post- BOTOX injections to investigate any structural changes.
Time Frame: 15-33 days between pre and post-Botox scans
Measure: Count of Participants; unit: Participants
Arm/Group | MRI Scans Pre and Post-Botox Injections
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 1-month
Arm/Group | Pre-Post
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03373162/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03373162/SAP_001.pdf